CLINICAL TRIAL: NCT03092388
Title: Evaluation Eines Leg Fluid Shift Und Erörterung Der hämodynamischen Und Respiratorischen Auswirkungen Auf Patienten Mit Chronischer Herzinsuffizienz Und Obstruktiver Oder Zentraler Schlafapnoe
Brief Title: Leg Fluid Shift in Patients With Chronic Heart Failure and Obstructive or Central Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Principal Investigator, Thomas Bitter, Senior Physician, Heart and Diabetes Center North-Rhine Westfalia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HDZNRW-KA_004_TB
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Obstructive Sleep Apnoea; Central Sleep Apnoea; Cheyne Stokes Respiration
Keywords: Sleep-Disordered Breathing; Heart Failure; Leg Fluid Shift
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea, Central; Cheyne-Stokes Respiration; Sleep Apnea Syndromes; Heart Failure | interventions — Polysomnography; Hemodynamic Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group Basic (Experimental): Patients receive Multi Frequency Bioimpedance Analysis (mfBIA) before and after sleep recording by Polysomnography/Polygraphy (PSG/PG) in hospital. Capillary Blood Gas Analysis (CBGA) is performed before and after sleep according to mfBIA.
  Interventions: Diagnostic Test: Multi Frequency Bioimpedance Analysis (mfBIA); Diagnostic Test: Polysomnography/Polygraphy (PSG/PG); Diagnostic Test: Capillary Blood Gas Analysis (CBGA)
- Study Group Extended (Experimental): Patients receive Multi Frequency Bioimpedance Analysis (mfBIA) before and after sleep recording by Polysomnography/Polygraphy (PSG/PG) in hospital. Capillary Blood Gas Analysis (CBGA) is performed before and after sleep according to mfBIA.
  Additionally, during daytime a special test with random parts of the study group basic is performed:
  A tilting table with hemodynamic monitoring is used to induce an artificial LFS by moving patients from vertical into horizontal position. Bodyfluid changes are monitored by mfBIA during this procedure.
  Interventions: Diagnostic Test: Multi Frequency Bioimpedance Analysis (mfBIA); Diagnostic Test: Polysomnography/Polygraphy (PSG/PG); Diagnostic Test: Capillary Blood Gas Analysis (CBGA); Diagnostic Test: Tilting Table with Hemodynamic Monitoring

INTERVENTIONS:
Diagnostic Test: Multi Frequency Bioimpedance Analysis (mfBIA) — Multi Frequency Bioimpedance Analysis (mfBIA) uses very small electric current at different frequencies (5, 50, 100 kHz) to measure the resistance and reactance of the entire body and different segmental body compartiments. With a special software total body fluid can be calculated. By analyzing raw data at different frequencies a detailed view on body and segments fluid distribution is possible.
  Other Names: Nutriguard M, Data Input, Darmstadt, Germany
Diagnostic Test: Polysomnography/Polygraphy (PSG/PG) — Sleep is digital recorded by using PSG/PG in hospital and manually analyzed by physicians according to current AASM guidelines.
Diagnostic Test: Capillary Blood Gas Analysis (CBGA) — CBGA is a less invasive method to gain arterial blood like gas samples without the punctation of an artery. After inducing a good capillary perfusion, capillary blood is taken by a small punctation of the tip of one ear. The sample is automatically analysed in a blood gas analyzer.
Diagnostic Test: Tilting Table with Hemodynamic Monitoring — A tilting table offers the opportunity to turn a study subject automatically from vertical into horizontal position and back. By using non-invasive monitoring technique, hemodynamic parameters are recorded permanently.
  Other Names: Task Force Monitor, CNsystems, Vienna, Austria
  Arms: Study Group Extended

SUMMARY:
This study aims to investigate the influence of a potential leg fluid shift (LFS) in patients with chronic heart failure (CHF) and obstructive sleep apnea (OSA) or central sleep apnea (CSA).

DETAILED DESCRIPTION:
Chronic heart failure (CHF) is a common disease in general western population with high levels of morbidity and mortality. Prospective risk factors need to be identified and investigated. The prevalence for sleep disordered breathing (SDB) in patients with CHF is higher compared to general population. Especially the occurence of CSA with its special breathing pattern of Cheyne-Stokes-Respiration (CSR) is frequent in CHF patients.The pathophysiology and relation inbetween sleep apnea (SA) and CHF isn´t completely identified yet. Multiple theories with different strategies try to explain the pathophysics and development of SA. Following one of these theories, patients with CHF often develop edema in lower body compartments. The idea is a possible influence of retrograde nocturnal LFS from lower body to upper body compartments which could induce pulmonal congestion. Therefore, an increased pulmonary capillary wedge pressure (PCWP) could irritate special pulmonal receptors resulting in CSR with periods of hyperventilation, related hypocapnia and central apnea events. OSA could be induced by fluid accumulation in the upper airway by retrograde fluid shift.

Patients with known CHF receive fluid measurements by b multi frequency bioimpedance analysis (mfBIA) the evening before and the morning after sleep is recorded using polygraphy (PG) or polysomnography (PSG) in hospital. Sleep results are analyzed by physicians using current guidelines of the American Academy of Sleep Medicine (AASM).

Capillary blood gas (CBG) samples are taken before and after sleep to examine the relation of fluid shift and blood gas changes.

A subgroup of the study group undergo additional investigation. Hemodynamic effects (e.g. reduced cardiac output (CO)) as a cause of a potential fluid shift is measured during wakefulness by using a tilting table. Hemodynamically relevant parameters are recorded non-invasively.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Heart Failure
* reduced left ventricular ejection fraction (LVEF) ≤ 45%
* NYHA I - IV

Exclusion Criteria:

* current existing sleep apnoea breathing therapy
* significant chronic obstructive pulmonary disease (COPD) Tiffenau-Index: <70%
* respiratory insufficiency with need for a long time oxygen therapy
* hypercapnic state in rest at day time
* acute myocardial infarction at moment of study
* instable angina pectoris at moment of study
* cardiac surgery in last twelve weeks
* stroke or TIA in last twelve weeks
* implantable cardioverter-defibrillator, if there is no security clearance of the fabricator
* chronic kidney disease > Stage III

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
∆ Leg Fluid Shift (LFS) | one night
  [%] Difference between the raw data of leg fluid volume before and after sleep.

SECONDARY OUTCOMES:
Apnea-Hypopnea-Index (AHI) | one night
  [/h], definition after current AASM guideline
Cheyne-Stokes-Respiration | one night
  [min] + [(%) of Total Sleep Time (TST)]
Oxygen-Desaturation-Index (ODI) | one night
  [/h], definition after current AASM guideline
Time Oxygen Saturation < 90% (TSpO2<90%) | one night
  [min] + [% (of TST)]
Oxygen Saturation (SpO2) | one night
Sleep Efficiency | one night
Longest Apnea time | one night
  [min]
Longest Hypopnea time | one night
  [min]
∆ partial pressure in capillary blood of carbon dioxide (pcCO2) | one night
  [mmHG] Difference of pcCO2 before and after sleep
∆ partial pressure in capillary blood of oxygen (pcO2) | one night
  [mmHG] Difference of pcO2 before and after sleep
∆ Resistance | one night
  [Ohm]
∆ Reactance | one night
  [Ohm]
∆ Total Body Water (TBW) | one night
  [l]
Blood Pressure (systolic, diastolic, mean) | one night
  [mmHg]

OTHER OUTCOMES:
Cardiac Index | one hour
  [(l/min)/m²] Cardiac output from left ventricle related to body surface during tilting table
∆ pcCO2 | one hour
  [mmHG] Difference of pcCO2 before and after tilting table
∆ pcO2 | one hour
  [mmHG] Difference of pcO2 before and after sleep
Thoracic Fluid Content (TFC) | one hour
  [1/kOhm]
∆ Leg Fluid Shift | one hour.
  [%] Difference between the raw data of leg fluid volume before and after tilting table.
∆ Total Body Water | one hour
  [l]
Oxygen Saturation | one hour
Blood Pressure (systolic, diastolic and mean) | one hour
  [mmHg]
∆ Resistance (legs, body) | one hour
  [Ohm] electrical resistance
∆ Reactance (legs, body) | one hour
  [Ohm] capacitive resitance

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bitter, MD, Study Director — Herz- und Diabeteszentrum NRW, Ruhr-Universitaet Bochum, Bad Oeynhausen, Germany; Schindhelm Florian, Principal Investigator — Herz- und Diabeteszentrum NRW, Ruhr-Universitaet Bochum, Bad Oeynhausen, Germany
Locations (1):
- Heart - and Diabetes CenteHerz- und Diabeteszentrum NRW, Ruhr-Universitaet Bochum, Bad Oeynhausen, Bad Oeynhausen, North - Rhine Westfalia, Germany

IPD SHARING:
Plan to Share IPD: No